CLINICAL TRIAL: NCT01769014
Title: In the Cantons Graubunden and Glarus as Well as in the Principality of Liechtenstein: Influence of Intensive Outpatient Treatment of People With Schizophrenia and Schizoaffective Disorder on Quality of Life and Adherence
Brief Title: Adherence and Quality of Life in People With Schizophrenia and Schizoaffective Disorder
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Psychiatrische Dienste Graubuenden (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2012-0178
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Quality of Life
Keywords: adherence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is the goal of this study adherence and quality of life in a population of people suffering from schizophrenia or schizoaffective disorder and to analyze if these factors are influenced by treatment, support, social services, and residential treatment. The study population is drawn from the the cantons Glarus and Graubunden as well as Liechtenstein.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder
* 18 - 65 years old
* treated in the PDGR within the past 19 years

Exclusion Criteria:

* organic brain disorder
* alcohol or drug dependence
* low intelligence
* unable to give consent
* no legal competency
* lacking knowledge of German language
* current psychiatric inpatient treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who suffer from schizophrenia or schizoaffective disorder, following DSM IV criteria and who live in the cantons Glarus, Graubuenden or the Principality of Liechtenstein.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Dienste Graubuenden, St. Moritz, Kanton Graubünden, Switzerland